CLINICAL TRIAL: NCT06893900
Title: Description of Care Pathways in Non-Traumatic Rotator Cuff Related Shoulder Pain Syndrome
Brief Title: Assessing Shoulder Pathways Involving the Cuff
Acronym: ASPIC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Conseil National de l'Ordre des Masseur Kinésithérapeutes (CNOMK) (Unknown); GIRCI Auvergne Rhône-Alpes (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-A01019-38
Record Dates: First submitted 2025-01-15; First posted 2025-03-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Rotator Cuff Shoulder Syndrome and Allied Disorders; Rotator Cuff Related Shoulder Pain
Keywords: rotator cuff; health economics; cost utility; incapacity; shoulder; non-traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary care non-traumatic shoulder pain: Patients will be enrolled if they receive care in France for non-traumatic shoulder disorder, that is related to the rotator cuff.

SUMMARY:
New recommendations regarding care pathways for the management of shoulder pain syndromes have recently been published. We aim to analyze and compare the existing care pathways and identify the most appropriate approaches for different patient profiles.

Our primary objective is to compare pain levels and shoulder function one year after your initial consultation with your general practitioner for this episode. We also seek to assess which healthcare professionals you consult for your shoulder management, the treatments you receive (e.g., analgesics), and any imaging studies you undergo (if prescribed).

We will send you notifications to remind you of the survey completion schedule and provide the link to access the questionnaire.

Participation in this study requires your commitment and adherence to the timeline, as missing data may compromise the analysis of results.

Non-participation in the study will not affect your current medical care.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff related shoulder pain
* Consultation with a general practitionner for this disorder in the 6 weeks prior to the inclusion

Exclusion Criteria:

* History of upper limb trauma associated with the current episode of shoulder pain
* Neurologic or rheumatismal shoulder disorder
* Frozen shoulder (current or past)
* History of advanced glenohumeral athritis
* History of shoulder surgery (on the affected side)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the French general population
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2027-03-27 (Estimated); Study Completion 2027-03-27 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain And Disability Index (SPADI) | 1 year
  The SPADI is a patient reported outcome measure assessing pain and function in the shoulder.

SECONDARY OUTCOMES:
Total number of different healthcare pathways and their description | 1 year
  Number and nature of different healthcare pathways that patients go through after having had a first general practitioner consultation for a first or new episode of non-traumatic rotator cuff related shoulder pain. E.g. : "surgical pathway", rheumatology pathway", "conservative pathway".
Number and proportion of patient in each healthcare pathway | 1 year
  Number and proportion of patient in each healthcare pathway that patients go through after having had a first general practitioner consultation for a first or new episode of non-traumatic rotator cuff related shoulder pain.
Delay for the first secondary care consultation | 1 year
  Delay between the GP referall and the consultation with a physiotherapist or a surgeon.
Number and nature of adverse event | 1 year
  Number and nature of adverse event in each pathway
Shoulder Pain And Disability Index (SPADI) | baseline, 2 weeks, 2, 4, 6 and 9 months
  Pain and function shoulder PROM
Pain Self-Efficacy Questionnaire-Fr | baseline, 6 and 12 months
  PROM assessing pain self-efficacy
Patient belief in the efficacy of rehabilitation | Baseline, 6 and 12 months
  Multiple choice question : "You believe that shoulder rehabilitation: 'allows for full recovery,' 'allows for partial recovery,' or 'does not allow for recovery.'"
Visual Analog Pain Scale | 1 year
  Self administered pain assessment
Tampa Scale of Kinesiophobia 11-item | Baseline and 6 and 12 months
  PROM assessing kinesiophobia
Fear and Avoidance Belief Questionnaire (FABQ) | baseline and 6 months
  PROM assessing fear and avoidance beliefs
EQ5D-5L | Baseline, 2, 4, 6, 9, 12 months
  PROM assessing quality of life
Direct costs | 2, 4, 6, 12 months
  Healthcare ressource consumption (Patient healthcare provider consultations, imaging, prescribed drugs, surgeries).
Indirect costs | 2, 4, 6 and 12 months
  Sick leaves
Referrals | 2, 4, 6, 9 and 12 months
  Number and types of referrals to other healthcare professionals
Patient satisfaction | 1 year
  Please respond to the statements below by circling the answer that best reflects your opinion regarding the care you received. (5 points likert scale for each item : Not at all satisfied - Not satisfied - Neutral - Satisfied - Completely satisfied and a Not Concerned option).
  The dimensions assessed are :
  1. Respect for my values, preferences, and needs
  2. Coordination and integration of the care I received
  3. Information, communication, and education about my condition
  4. Physical comfort during care
  5. Emotional support, relief of my fears and anxiety
  6. Involvement of my family and close relatives in my care
  7. Transition and continuity of care
  8. Accessibility of care
Patient preferences and motivation regarding a surgical or conservative pathway | baseline, 2, 4, 6, 9 and 12 months
  Semi-guided interviews with patients from each identified pathway at different points in time.
Dominant upper limb and involved upper limb | Baseline
  Dominant upper limb: left, right, or neither Affected upper limb: left, right, or both
Quick DASH | At baseline and 12 months
  The sort version of the "disability of the arm, the shoulder and the hand" patient reported outcome measure.
PASS | 12 months
  Patient Acceptable Symptom State : "Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?" - Dichotomic answer.
Anchor-based MCID | Baseline, 2, 4, 6, 9 and 12 months
  Patients are asked : "Since the last questionnaire, my shoulder pain and function has :
  * Significantly improved
  * Improved, but not really changed
  * Neither improved nor deteriorated
  * Worsened, but not really changed
  * Significantly worsened"

CONTACTS AND LOCATIONS:
Overall Officials: Thomas LATHIERE, PT, PhDc, Principal Investigator — Grenoble Alpes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided